CLINICAL TRIAL: NCT04501055
Title: A Prospective Multicenter Randomized Controlled Trial Assessing Whether the Perineal Nerve Block Approach is Better Than the Periprostatic Block for the Pain Control in Men Who Undergo Transperineal Prostate Biopsy
Brief Title: Anesthesia in PROstate Biopsy Pain Obstruction Study
Acronym: APROPOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shi Shi Municipal General Hospital (Unknown); People's Hospital of Yiyuan County (Unknown); The First Affiliated Hospital of University of Science and Technology of China (Other); Guang'an people's hospital of Sichuan province (Other); Chinese University of Hong Kong (Other); Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APROPOS-01
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; transperineal prostate biopsy; perineal nerve block; periprostatic block; anesthesia
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, the investigator and the outcomes assessor were all masked. Only the care provider who performed the anaesthesia were not blinded but they were not involved in the subsequent prostate biopsy, pain assessment, data collection and data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineal nerve block (Experimental): Man receive the perineal nerve block before under the transperineal prostate biopsy
  Interventions: Behavioral: perineal nerve block
- Periprostatic block (Active Comparator): Man receive the periprostatic block before under the transperineal prostate biopsy
  Interventions: Behavioral: periprostatic block

INTERVENTIONS:
Behavioral: perineal nerve block — An anesthesia method to block perineal nerve
  Arms: Perineal nerve block
Behavioral: periprostatic block — An anesthesia method to block periprostate
  Arms: Periprostatic block

SUMMARY:
This is a multicentre randomized controlled trial in comparison of the perineal nerve block approach between the periprostatic block in the pain control in men undergo a transperineal prostate biopsy.

DETAILED DESCRIPTION:
This trial is a prospective, multicentre, randomized controlled study in which all men plan to undergo a transperineal prostate biopsy. This study aims to determine whether the perineal nerve block approach is better than the periprostatic block in the pain control in men undergo a transperineal prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 80 years old
2. a PSA level of 4 - 20 ng/ml, and/or suspicious rectal examination findings;
3. fully understand the clinical trial protocol and sign the informed consent;

Exclusion Criteria:

1. local anesthetic allergy patients;
2. symptomatic acute or chronic inflammation of the prostate;
3. cannot tolerate prostate biopsy or has contraindication to biopsy;
4. patients judged by the investigator to be unsuitable to participate in the clinical trial;

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
The pain of the biopsy procedure | within10 minutes after the prostate biopsy
  The pain will be measured by numerical rating scale（NRS), which distributed from 0 to 10. 0 represents no pain, and 10 represents the worst pain imaginable.

SECONDARY OUTCOMES:
The pain in 1,6, and 12 hours after the biopsy | 1,6, and 12 hours after the biopsy
  The pain in 1,6, and 12 hours will be measured by numerical rating scale（NRS), which distributed from 0 to 10. 0 represents no pain, and 10 represents the worst pain imaginable.
Changes in blood pressure during biopsy procedure | During the biopsy procedure
  The changes will be measured and recorded by multi-parameter monitoring
Changes in heart rate during biopsy procedure | During the biopsy procedure
  The changes will be measured and recorded by multi-parameter monitoring
Changes in breath rate during biopsy procedure | During the biopsy procedure
  The changes will be measured and recorded by multi-parameter monitoring
The detection rate for prostate cancer | within 1 month after the biopsy
  The detection rate for any of the prostate cancer
The detection rate for clinically significant prostate cancer | within 1 month after the biopsy
  The detection rate for prostate cancer with a ISUP>2
External manifestation of pain | 10 minutes within biopsy
  A questionnaire with five items: the degree of facial expression (0 for no particular expression or smile; 1 for an occasional grimace or frown, a withdrawn expression, or a disinterested expression; 2 for frequent or constant quivering chin or a clenched jaw), the degree of activity (0 for lying quietly or being in a normal position, 1 for slight contractions of the hip muscles or slight movements of hip, 2 for severe contractions of the hip or lifting the hip out of the bed), the degree of voice expression (0 for quiet or normal communication, 1 for an occasional moan or weeping sound, 2 for constant moaning or sobbing and screaming), the degree of pacification (0 for being peaceful and not requiring pacification, 1 for being able to be comforted easily, 2 for being difficult to comfort) and the degree of cooperation (0 for being calm and cooperative, 1 for language resistance, 2 for body resistance).
Anaesthesia satisfaction | 24 hours after the biopsy
  A questionnaire with five items :whether the pain during the biopsy was less severe than expected (scores from 0 to 10, where 0 represents far less severe and 10 represents far more severe than expected); whether the pain after anaesthesia was less severe than the pain during anaesthesia (scores from 0 to 10, where 0 represents far less severe and 10 represents far more severe); weather the patient is satisfied with the overall feeling of the biopsy (scores from 0 to 10, where 0 represents the highest level of satisfaction and 10 represents the lowest level of satisfaction); whether the patient would recommend this type of biopsy to other patients (scores from 0 to 10, where 0 represents they would highly recommend it and 10 represents they would definitely not recommend it); and whether the patient would still want to choose this way if they have to undergo another biopsy (scores from 0 to 10, where 0 represents very willing to choose it and 10 represents extreme reluctance).
Adverse event | Within 1 week after the biopsy
  Any of the adverse events during the trial
The number of biopsy cores | 10 minutes within biopsy
  The number of biopsy cores
The location of each biopsy core | 10 minutes within biopsy
  The location of each biopsy core
Prostate volume | within 3 months before the biopsy procedure
  The prostate volume will be measured by MRI before biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wang, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Once available, the results of this trial will be disseminated to an international peer-reviewed journal and presentations at international or national academic conferences. The data will be made available upon request to researchers a) who provide a methodologically sound proposal and b) whose proposed use of the data has been approved by an independent ethical review committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after publication with no end date

REFERENCES:
- [Derived] He BM, Ka-Fung Chiu P, Tao T, Lan JH, Cai JT, Zhou SC, Li RB, Ren Y, Ka-Lun LO, Xu RY, Chen JR, Lan D, Gao JL, Chu SG, Jin ZC, Huang FF, Shi ZK, Yang QW, Zhou H, Wang SD, Ji TR, Han QP, Wang CM, Chi-Fai NG, Wang HF; APROPOS Group. Perineal nerve block versus periprostatic block for patients undergoing transperineal prostate biopsy (APROPOS): a prospective, multicentre, randomised controlled study. EClinicalMedicine. 2023 Mar 23;58:101919. doi: 10.1016/j.eclinm.2023.101919. eCollection 2023 Apr. PMID 37007736
- [Derived] He BM, Li RB, Wang HF. Anaesthesia in PROstate Biopsy Pain Obstruction Study: A Study Protocol for a Multicentre Randomised Controlled Study Evaluating the Efficacy of Perineal Nerve Block in Controlling Pain in Patients Undergoing Transperineal Prostate Biopsy. Front Surg. 2021 Oct 6;8:649822. doi: 10.3389/fsurg.2021.649822. eCollection 2021. PMID 34692757